CLINICAL TRIAL: NCT02127151
Title: A Single Arm Phase II Trial of BMN 673 for Inoperable, Advanced Endometrial Cancer With Retrospective PTEN, MSI and MRE11 Analysis
Brief Title: A Parp Inhibitor (BMN 673) for Inoperable Advanced eNDometrial cAncer
Acronym: PANDA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of Industry support for the study
Sponsor: University College, London (Other)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/13/0045; 2013-003469-32 (EudraCT Number)
Record Dates: First submitted 2014-04-14; First posted 2014-04-30 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMN 673 (Experimental): BMN 673 daily until progression, death, unacceptable toxicity, withdrawal of consent or any other criterion felt by the Investigator to preclude continuation of treatment.
  Interventions: Drug: BMN 673

INTERVENTIONS:
Drug: BMN 673 — Starting oral dose of 1.0 mg once daily to be taken until progression, death, unacceptable toxicity, withdrawal consent or any other criterion felt by the Investigator to preclude continuation of treatment.

SUMMARY:
A Single Arm Phase II Trial of BMN 673 for Inoperable, Advanced Endometrial Cancer With Retrospective PTEN, MSI and MRE11 Analysis

PTEN= Phosphatase and tensin homolog MSI= Microsatellite instability MRE11= Double-strand break repair protein MRE11A

This trial will investigate whether the drug BMN 673 has therapeutic benefit in the treatment of advanced endometrial cancer. Nearly 8,000 patients are diagnosed with endometrial cancer in the UK every year. A significant proportion are either diagnosed with advanced disease which may be inoperable and/or metastatic (i.e spread to other organs outside the endometrium), or curable disease which relapses following first line treatment. There is no established standard of care for these patients as both chemo and hormone therapy has limited effectiveness and survival benefit. Survival rates have not improved in the past 20 years. Furthermore there are no so called 'targeted' drugs licensed for its treatment i.e. drugs that block the growth and spread of cancer by interfering with specific molecules involved in tumor growth and progression. This leaves an unmet need for effective systemic treatments for advanced, inoperable and metastatic endometrial cancer.

BMN 673 has been shown to be potentially effective in treating cancers known to behave similarly to endometrial disease, both in the laboratory and in Phase I studies involving patients with advanced cancers. Similarly the drug appears to be relatively tolerable. A Phase II trial such as the one proposed by this application could demonstrate activity that might lead to a new effective treatment for patients with inoperable, advanced, recurrent or metastatic endometrial cancer, while the proposed substudy also presents the possibility of discovering a subset of patients more likely to derive benefit from BMN 673.

This trial is for adult women (18 and above) with advanced, inoperable or metastatic endometrial cancer. Patients will be recruited from approximately 15 National Health Service (NHS) Trusts based in the United Kingdom (UK). The study is expected to last approximately 18-24 months in terms of recruitment time, and a maximum of 100 eligible women will be registered. All patients will receive BMN 673 until their disease worsens or their doctor decides they should stop treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically confirmed endometrial cancer. All histological subtypes except for carcinosarcoma are eligible
* Evidence of inoperable, advanced, recurrent or metastatic disease by imaging and/or histological criteria
* ≤ 1 previous line of systemic cancer therapy for inoperable, advanced, recurrent or metastatic endometrial cancer. Chemotherapy in the adjuvant setting is not considered a prior line of therapy unless recurrence occurred during adjuvant treatment or ≤ 6 months after the last treatment; first line treatment of advanced disease must include at least one cytotoxic agent to be considered as a line of therapy; prior hormonal treatment is not considered a line of therapy in any setting
* Written informed consent obtained prior to any screening procedures
* Patients must give consent for provision of archival histological tissue for the purposes of translational research. If archival tissue is not available or is of insufficient quantity and/or quality, the patient will have the option to consent to undergo biopsy where feasible. If biopsy is not feasible or the patient does not give consent for biopsy when archival tissue is not available, the patient will not be eligible for the trial. The quality and quantity of archival tissue will be assessed by a suitably qualified individual, usually a histopathologist, at site to ensure adequate tissue sample available for testing PTEN, MSI and MRE11
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-2
* Life expectancy ≥ 12 weeks
* Patient has at least one site of measurable disease on radiological imaging (i.e. target lesion) as per RECIST v1.1
* Evidence of non-childbearing status and must not be lactating OR must have postmenopausal status
* Adequate bone marrow and organ function

Exclusion Criteria:

* Prior treatment with a poly adenosine diphosphate ribose polymerase (PARP) inhibitor
* Progressive disease ≤ 3 months after platinum-based chemotherapy
* Active uncontrolled infection including known Hepatitis B, Hepatitis C or HIV
* Obstruction of the gastrointestinal tract or other reason preventing effective oral administration of medication
* Serious concomitant non-malignant disease, uncontrolled organ dysfunction or medical disorder considered by the Investigator to make the subject unsuitable for trial participation including any psychiatric disorder that prevents informed consent
* Significant active cardiovascular disease
* Symptomatic brain metastases
* Immunosuppressant therapy or considered to be otherwise immunocompromised
* Myelodysplastic syndrome/acute myeloid leukaemia
* Major surgery ≤ 28 days prior to registration, or ongoing clinically significant post-surgical complications
* Chemotherapy, radiotherapy (a single fraction of palliative radiotherapy is allowed provided that the site being treated is not subsequently used as a target lesion as per RECIST v1.1 for the purpose of assessing tumour response on trial), immunotherapy or other investigational therapy for cancer ≤ 21 days prior to registration (42 days for nitrosoureas, mitomycin-C)
* Unresolved clinically significant toxicities from prior systemic therapy
* Known hypersensitivity to any of the agents or excipients to be administered
* Unwillingness or inability to comply with the trial protocol
* Patients with a history of other malignancy ≤ 3 years prior to registration with the exceptions of a) cone-biopsied in situ carcinoma of the cervix uteri; b) basal or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) rate | 6 months
  Measured from date of first BMN 673 dose to first progression (defined using Response Evaluation Criteria in Solid Tumours (RECIST) v1.1) or death, whichever is the sooner.

SECONDARY OUTCOMES:
Best Response | Up to 30 months
  Measured from the date of first BMN 673 dose.
Overall survival (OS) | Up to 30 months
Response at each radiological assessment | Up to 30 months
Duration of Response (DoR) | Up to 30 months
Median PFS | Up to 30 months
Safety and toxicity | Up to 30 months
  Common Terminology Criteria for Adverse Events (CTCAE) v4.03 grade 3-4 toxicity; dose reductions, omissions, delays; exposure; compliance.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kristeleit, Principal Investigator — University College, London
Locations (16):
- United Kingdom (16):
  - Royal Sussex County Hospital, Brighton, East Sussex
  - The Beatson West of Scotland Cancer Centre, Glasgow, Greater Glasgow
  - St Bartholomew's Hospital, London, Greater London
  - University College Hospital, London, Greater London
  - The Christie Hospital, Manchester, Greater Manchester
  - Western General Hospital, Edinburgh, Lothian
  - The Churchill Hospital, Oxford, Oxfordshire
  - Velindre Cancer Centre, Cardiff, South Glamorgan
  - St James's University Hospital, Leeds, South Yorkshire
  - Royal Marsden Hospital (Sutton), Sutton, Surrey
  - The Clatterbridge Cancer Centre, Bebington, Wirral
  - Bristol Haematology and Oncology Centre, Bristol
  - East Kent Hospitals University NHS Foundation Trust, Kent
  - Guy's Hospital, London
  - The Royal Marsden Hospital (London and Surrey), London and Surrey
  - Northern Centre for Cancer Care, Newcastle

REFERENCES:
- See also: Trial page on the University College London (UCL) Cancer Trials Centre website — http://www.ctc.ucl.ac.uk/TrialDetails.aspx?TrialID=79&TrialName=PANDA